CLINICAL TRIAL: NCT01053325
Title: A Clinical Trial to Establish The Effectiveness of Daily Co-trimoxazole Prophylaxis For Prevention of Malaria in Pregnancy
Brief Title: Establishing Effectiveness of Daily Co-trimoxazole Prophylaxis For Prevention of Malaria in Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Tropical Diseases Research Centre, Zambia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ITMP0409
Record Dates: First submitted 2010-01-18; First posted 2010-01-21 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Malaria in Pregnancy; HIV Infections
Keywords: Malaria; Pregnancy; Prevention; HIV; Sub-Sahara Africa
MeSH Terms: conditions — HIV Infections; Malaria | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- CTX in HIV-negative women (Experimental): CTX daily prophylaxis in HIV-negative pregnant women
  Interventions: Drug: Cotrimoxazole prophylaxis
- CTX in HIV-positive women (Experimental): CTX daily prophylaxis in pregnant women who are infected with HIV
  Interventions: Drug: Cotrimoxazole prophylaxis
- SP IPT in HIV-negative women (Active Comparator): Intermittent Preventive Treatment with SP in HIV-negative pregnant women
  Interventions: Drug: SP IPT
- IPT SP in HIV-positive women (Active Comparator): Intermittent Preventive Treatment with SP in HIV-positive pregnant women
  Interventions: Drug: SP IPT
- CTX in HIV-positive pregnant women with CD4<350 (Active Comparator): Daily prophylaxis with cotrimoxazole in HIV-positive pregnant women with CD4<350
  Interventions: Drug: Cotrimoxazole prophylaxis

INTERVENTIONS:
Drug: Cotrimoxazole prophylaxis — Daily prophylaxis with cotrimoxazole
  Other Names: CTX; Bacrtim (R)
  Arms: CTX in HIV-negative women; CTX in HIV-positive pregnant women with CD4<350; CTX in HIV-positive women
Drug: SP IPT — Intermittent preventive treatment with sulphadoxine-pyrimethamine
  Other Names: SP; Fansidar (R)
  Arms: IPT SP in HIV-positive women; SP IPT in HIV-negative women

SUMMARY:
Malaria is a major contributor of disease burden in Sub-Saharan Africa: 90% of global cases occur there, and pregnant women and children under 5 years are the most vulnerable. Malaria in pregnancy increases risks of abortion, stillbirth, prematurity, intrauterine growth retardation and maternal anemia, and is associated with higher risk of low birth weight and perinatal, neonatal and infant mortality. For prevention and control of malaria in pregnancy, the WHO recommends Intermittent Preventive Treatment (IPT) with antimalarial drugs, insecticide treated nets (ITNs) and effective treatment of malaria and anemia.

HIV in pregnancy increases the risks of malaria, and it seems that the efficacy of IPT with the drug sulphadoxine-pyrimethamine (SP) is decreased in HIV+ pregnant women.

Malaria prevention in pregnancy in Zambia relies on ITNs and IPT with SP. Daily prophylaxis with cotrimoxazole (CTX) effectively reduces mortality and morbidity in HIV+ individuals, and antibiotic therapy during pregnancy might help to decrease adverse pregnancy outcomes. CTX prophylaxis improves birth outcomes in HIV+ women with CD4<200/µl: a study concluded that antenatal provision of CTX was beneficial for HIV+ pregnant women with low CD4 but not in women with ≥200/µl (however, this study was carried out in an area with very low risk of malaria , and CTX may have a different effect depending on endemic conditions). The WHO recommends daily CTX in addition to ARVs, to prevent opportunistic infections in all HIV+ patients.

Concurrent administration of SP and CTX may increase the incidence of severe adverse reactions in HIV+ patients, so WHO has promoted CTX prophylaxis as an alternative to SP for the IPT in immuno-compromised pregnant women. Unfortunately, there is insufficient information on the effectiveness of daily CTX for preventing malaria infection in pregnancy: so, SP is still the only antimalarial recommended by WHO for this purpose. With the increase in SP resistance and with the newer antimalarials still being studied for safety and efficacy in pregnancy, CTX could be an alternative for SP in reducing malaria and malaria-related morbidity and mortality in pregnancy.

This study will try to to see if in HIV- and HIV+ pregnant women, CTX is not inferior to SP in reducing placental parasitaemia. Such information is needed to issue updated, effective guidelines on malaria prevention in pregnancy

DETAILED DESCRIPTION:
Malaria is a major contributor of the disease burden in Sub-Saharan Africa: some 90% of global cases occur in Sub-Saharan Africa, with pregnant women and children < 5 representing the most vulnerable population. P.falciparum infection in pregnancy leads to parasite sequestration in the maternal placental vascular space, causing increased risks of abortion, stillbirth, prematurity, intrauterine growth retardation and maternal anaemia; it is also associated with increased risk of low birth weight (LBW) and perinatal, neonatal and infant mortality.In low transmission areas, malaria can be severe with a high risk of maternal and perinatal mortality (up to 60-70%). In highly endemic areas, malaria is still associated with maternal anaemia, LBW and stillbirth. For prevention and control of malaria in pregnancy, the WHO recommends Intermittent Preventive Treatment (IPT), insecticide treated nets (ITNs) and effective case management for malaria and anaemia.

HIV-1 infection in pregnancy increases the risks of malaria. In HIV+ pregnant women, in addition, the efficacy of IPT with sulphadoxine-pyrimethamine (SP) appears decreased.

In Zambia, the malaria incidence rate increased from 121.5/1000 in 1976 to 482.0/1000 in 2003. The high rates were predominantly evident among pregnant women and children <five. Malaria prevention in pregnancy in Zambia relies on ITNs and IPT with SP.

Several studies in Zambia and Uganda demonstrated that daily cotrimoxazole (CTX) prophylaxis is effective in reducing mortality and morbidity in HIV+ individuals and that antibiotic therapy during pregnancy might impact positively to the reduction of adverse pregnancy outcomes. CTX prophylaxis significantly improves birth outcomes in HIV+ women with CD4<200/µl. A recent study in Zambia concluded that antenatal provision of CTX was beneficial for HIV+ pregnant women with low CD4 but not in women with ≥200/µl. However, this study was carried out in an area with an extremely low risk of malaria infection; CTX may have had a different impact if malaria transmission was either holo or hyperendemic. Today, WHO recommends daily CTX in addition to ARVs, to prevent opportunistic infections in HIV+, regardless of the background prevalence of CTX microbial resistance.

Concurrent administration of SP and CTX has been associated with increased incidence of severe adverse reactions in HIV+ patients. Therefore, WHO has promoted CTX prophylaxis as an alternative to SP for the IPT in immuno-compromised (CD4 < 350/µl)pregnant women. Unfortunately, there is insufficient information on the effectiveness of daily CTX for preventing malaria infection (placental parasitaemia) and its consequences (maternal anaemia and low birth weight) in pregnancy: so, presently, SP is the only antimalarial treatment for which data on efficacy and safety for IPT is available, and the WHO recommends that at least 2 doses of SP are given after the first trimester. With the documented increase in SP resistance and with the newer antimalarials still being studied for safety and efficacy in pregnancy, CTX could be an alternative for SP in reducing malaria and malaria related morbidity and mortality in pregnancy.

The focus of this study is the malaria related outcome in pregnancy: we will target both HIV negative and HIV positive pregnant women, assuming that CTX is not inferior to SP in reducing placental parasitaemia. Such information is urgently needed in order to issue updated, effective guidelines on intermittent preventive treatment in pregnant women.

An open label clinical trial is the best design to assess the research question and its consequences on the offspring, both in HIV negative pregnant women and in HIV positive pregnant women with CD4 count ≥350/µl. The parallel design was chosen evaluate to each group separately, as HIV might interact with CTX efficacy. Offsets for efficacy were based on literature review.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pregnancy (through palpable fundus and/ or positive pregnancy test)
* Gestational age between 16 and 28 weeks
* Hb > 7 g/dl, by Hemocue
* No symptoms consistent with malaria
* Residence within the health facility catchment's area
* Willingness to deliver at the health facility
* Willingness to adhere to all requirements of the study (including HIV-1 voluntary counselling and testing)
* Ability to provide written informed consent. If the woman is a minor of age/not emancipated, the consent must be given by a parent or legal guardian according to national law (however, in this case, also the minor woman will sign the consent form, to document that she is freely giving her assent to take part in the study).

Exclusion Criteria:

* History of allergy to study drugs, or previous history of allergy to sulpha drugs
* History or presence of major illnesses likely to influence pregnancy outcome including diabetes mellitus, severe renal or heart disease, or active tuberculosis
* Any significant illness at the time of screening that requires hospitalization
* Intent to move out of the study's catchment area before delivery or deliver at relative's home out of the catchment's area;
* Prior enrolment in the study or concurrent enrolment in another study
* Severe anaemia (Hb<7 g/dl)
* Previous history of unfavourable pregnancy outcome: pre-eclampsia, caesarean section, stillbirth.
* Eligible HIV-positive women who, following the National guidelines, have to be put on CTX prophylaxis (e.g. having a CD4 count <350/µl) or already on CTX and/or ARV treatment will be excluded from the RCT but included in a prospective observational cohort and receive 2 tablets of CTX daily

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 848 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To establish that in HIV negative pregnant women co-trimoxazole prophylaxis is non inferior to SP IPT with respect to birth weight at delivery (or within 24 hours). Non inferiority is defined as a difference in mean birth weights of no more than 100g. | Up to the end of pregancy

SECONDARY OUTCOMES:
To evaluate the effectiveness of co-trimoxazole prophylaxis and SP IPT in reducing placenta malaria in HIV+ pregnant women with CD4 ≥ 350/µl and in the combined group of HIV- and HIV+ pregnant women with CD4 ≥ 350/µl | Up to the end of pregnancy
To evaluate the effectiveness of CTX and SP IPT in reducing malaria peripheral infection, in HIV negative, and in HIV positive pregnant women with a CD4 cell count ≥ 350/µl | Up to the end of pregnancy
To evaluate the effect of CTX and SP IPT on the offspring by measuring the gestational age at delivery, perinatal mortality and birth weight, in HIV negative pregnant women and in HIV positive pregnant women with a CD4 cell count ≥ 350/µl | At delivery
To compare the effectiveness and safety profiles of CTX prophylaxis to that of SP IPT, in HIV negative pregnant women and in HIV positive pregnant women with a CD4 cell count ≥ 350/µl | Up to the end of pregancy

CONTACTS AND LOCATIONS:
Overall Officials: Christine Manyando, MD, Principal Investigator — Tropical Diseases Research Centre, Zambia; Umberto D'Alessandro, MD, PhD, Study Director — Insitute of Tropical Medicine, Antwerp, Belgium
Locations (1):
- Kabuta Health Centre, Kabuta, Nchelenge District, Luapula Province of, Zambia